CLINICAL TRIAL: NCT01530282
Title: Non-invasive Respiratory Mechanics Assessment During Spontaneous / Assisted Breathing: The ERNI (Elastance, Resistance, Non Invasive Measurements) Study
Brief Title: Non-invasive Measurements of Elastance and Resistance
Acronym: ERNI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Ranieri, MD Professor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ERNI-0073496
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory Insufficiency [C08.618.846]
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- measurement of respiratory mechanics (Experimental): Invasive method: two catheters will be inserted to measure reference respiratory mechanics Non_invasive method: airway pressure measured during a 150-200 ms occlusion at the beginning of inspiration.
  Interventions: Other: Invasive method; Other: Non invasive method

INTERVENTIONS:
Other: Invasive method — Esophageal and gastric catheters to measure respiratory mechanics (static and dynamic)
Other: Non invasive method — Non_invasive method: airway pressure measured during a 150-200 ms at the beginning of inspiration

SUMMARY:
The study aims to assess the agreement between respiratory mechanics parameters measured noninvasively by means of brief airways occlusions at the beginning of inspiration and the reference parameters obtained with standard techniques of esophageal and gastric pressure under static and dynamic conditions in a mixed population of ICU patients mechanically ventilated in pressure support ventilation mode.

ELIGIBILITY:
Inclusion Criteria:

* intact respiratory drive;
* PaO2/FiO2 ratio > 150 with a positive end-expiratory pressure (PEEP) ≤ 8 cmH2O;
* pH between 7.35 and 7.45;
* patient alert, conscious, and cooperative with a Glasgow Coma Scale ≥ 10.

Exclusion Criteria:

* infection, sepsis or septic shock; (with fever no)
* hemodynamic instability;
* respiratory centres depression;
* esophageal deformity, or gastric/esophageal illnesses;
* previous recent gastric/esophageal surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Non-invasive respiratory mechanics measurement | 2 hours
  use of 150-200 ms airway occlusions at the beginning of inspiration to measure non-invasive respiratory mechanics

CONTACTS AND LOCATIONS:
Overall Officials: Vito Marco VM RANIERI, MD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine, University of Turin, Italy